CLINICAL TRIAL: NCT04839861
Title: Examining the Impacts of Parent-Child Interactive Activities as an Adjunct to Mightier Play
Brief Title: Examining the Impacts of Parent-Child Interactive Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromotion Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 874MIGH21
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Emotional Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mightier Online Games (Active Comparator): 6 weeks of use ad-libitum. Parents will be encouraged to have their children play Mightier online games at least 3 times a week for the 6 week duration.
  Interventions: Behavioral: Mightier online gameplay
- Mightier Online Plus Offline Family Games (Experimental): 6 weeks of use ad-libitum. Parents will be encouraged to have their children play Mightier online games at least 3 times a week for the 6 week duration. Parents will be encouraged to play Mightier offline Family Games at least once a week for the 6 week duration.
  Interventions: Behavioral: Mightier Family Games; Behavioral: Mightier online gameplay

INTERVENTIONS:
Behavioral: Mightier Family Games — Mightier Family Games includes five offline card games that can be played by two or more people. During card game play, one player wears the Mightier heart rate monitor, and can see a representation of their heart rate on a separate screen within the Mightier app. Each game includes elements that are tied to heart rate.
  Arms: Mightier Online Plus Offline Family Games
Behavioral: Mightier online gameplay — Mightier is a video-game-based biofeedback intervention that capitalizes on children's love of video games to increase emotional awareness and facilitate emotion regulation practice through heart rate (HR) control. Each family receives a Mightier Kit (Mighty Band heart rate monitor, dedicated Mightier tablet unless the family prefers to use their own device) and the Mightier App. Children wear a "Mighty Band" heart rate monitor on their arm while they play any one of 26+ games. As their heart rate rises the games become more difficult. For example, during a cooking game, smoke may appear on the screen and obscure the player's view. Children can either opt into an explicit cool down activity (deep breathing, progressive muscle relaxation, crossing the midline, or visualization) or cool down on their own.
  Other Names: Mightier

SUMMARY:
The purpose of this study is to demonstrate the effects of online and offline play of games on the Mightier game platform, in comparison to the effects of Mightier online play alone.

DETAILED DESCRIPTION:
Mightier is a mobile app-based biofeedback video game platform that facilitates emotion regulation skill-building among children ages 6-14. The technology behind Mightier's mobile app has been validated in two independent sham-controlled randomized controlled trials, where the investigators have seen decreases in clinical symptoms of aggression and disruptive behaviors, as well as lowered family stress without adverse events.

Mightier will soon introduce offline Mightier Family Games to its product line. Mightier Family Games will include offline, interactive components that have not previously been incorporated into Mightier play. Studies have shown that improvements in child behavior and child-parent relationships are among the many benefits of family play.

For the proposed study, families with no prior Mightier exposure will engage in different types of Mightier play for six weeks, to demonstrate the effects of online and offline Mightier play in comparison to the effects of Mightier online play alone. Mightier will recruit families through social media, then Mightier will randomly assign participants to one of two groups: a Mightier online play only group, and a Mightier online and offline play group. The investigators will aim to enroll 20 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 at the time of screening
* Regular access to WiFi (for Mightier gameplay device connection)

Exclusion Criteria:

* Prior Mightier use
* Diagnosed Intellectual Disability (by history)
* Planned medication changes during the 6-week study period

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Change in child irritability from baseline measured on ARI-P at Week 7 | Baseline and Week 7
  Affective Reactivity Index-Parent Report (ARI-P): The ARI is a 7-item scale that consists of 6 symptom items and 1 impairment item. The scale was designed to determine irritable mood rather than behavioral consequences such as hostility and acts of aggression (Stringaris et al., 2012). The individual items are scored 0,1, 2, and only the first six items are summed to form the total score, with a minimum score of 0 and a maximum score of 18, and higher scores indicating greater severity of irritability symptoms. The seventh item is an impairment item and it is analysed separately, with a minimum score of 0 and a maximum score of 3, and higher scores indicating greater irritability symptom severity.
Change in child-parent relationship from baseline measured on CPRS-SF at Week 7 | Baseline and Week 7
  Child-Parent Relationship Scale (CPRS-SF): The CPRS-SF is a 15- item The CPRS (Pianta, 1992) is a self-report instrument completed by parents that assesses their perceptions of their relationship with their child. The 15 items are rated on 5-point Likert scales. It is applicable to children ages 3-12. The CPRS-SF is scored in two subscales: an 8-item Conflict subscale (minimum score = 8, maximum score = 40, higher score indicates greater conflict), and a 7-item Closeness subscale (minimum score = 7, maximum score = 35, with greater score indicating greater closeness).
Parent perception of change in child emotion regulation from baseline measured on GIS at Week 7 | Week 7
  Global Improvement Scale (GIS): The GIS is a parent self-report question that asks parents if they have noticed any overall improvements in their child's emotion regulation, with response options ranging from (1) very much improved to (7) very much worse. Minimum score = 1, Maximum score = 7, with higher numbers indicating less improvement, or worsening. The GIS has not been scientifically validated.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kahn, PhD, Principal Investigator — Neuromotion Labs Inc
Locations (1):
- Neuromotion Labs, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Only Mightier research staff will have access to individual participant data, including family demographics data and data from parent self-report measures.

REFERENCES:
- [Background] Stringaris A, Goodman R, Ferdinando S, Razdan V, Muhrer E, Leibenluft E, Brotman MA. The Affective Reactivity Index: a concise irritability scale for clinical and research settings. J Child Psychol Psychiatry. 2012 Nov;53(11):1109-17. doi: 10.1111/j.1469-7610.2012.02561.x. Epub 2012 May 10. PMID 22574736
- [Background] RC Pianta - Unpublished measure, University of Virginia, 1992